CLINICAL TRIAL: NCT05115630
Title: A Phase I/II Clinical Trial of "Off-the-shelf" NK Cell Administration in Combination With Allogeneic SCT to Decrease Disease Relapse in Patients With High-risk Myeloid Malignancies Undergoing Matched Related, Matched Unrelated, One Antigen Mismatched Unrelated, or Haploidentical Stem-cell Transplantation
Brief Title: Off-the-shelf NK Cells + SCT for Myeloid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0329; NCI-2021-12094 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-10-11; First posted 2021-11-10 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Myeloid Malignancies; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Cyclophosphamide; Mesna; Filgrastim; Melphalan; fludarabine phosphate; Tacrolimus; Mycophenolic Acid; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cyclophosphamide (Experimental): On Days 3 and 4, you will receive cyclophosphamide by vein over about 3 hours to help lower the risk of graft-versus-host disease
  Interventions: Drug: Cyclophosphamide
- Mesna (Experimental): On Days 3 and 4, You will also receive mesna by vein over 30 minutes every 4 hours for a total of 10 mesna doses.
  Interventions: Drug: Mesna
- Filgrastim (Experimental): Starting on Day 7, you will begin to receive filgrastim as an injection under the skin 1 time a day.
  Interventions: Drug: Filgrastim
- Melphalan (Experimental): On Day -7, you will receive melphalan by vein over about 30 minutes.
  Interventions: Drug: Melphalan
- Fludarabine phosphate (Experimental): On Days -7, -6, -5, and -4, you will receive fludarabine by vein about 1 hour.
  Interventions: Drug: Fludarabine phosphate
- Tacrolimus (Experimental): Starting on Day 5, you will begin receiving tacrolimus to help lower the risk of GVHD. You will begin by receiving it nonstop by vein until you are able to take it by mouth. You will then take tacrolimus by mouth 2 times a day for about 3 months.
  Interventions: Drug: Tacrolimus
- Mycophenolate mofetil (Experimental): by mouth 3 times a day for 90 days or longer.
  Interventions: Drug: Mycophenolate mofetil
- Total Body Irradiation One Dose (Experimental): on Day -2, you may receive 1 dose of total body irradiation (TBI).
  Interventions: Drug: Total Body Irradiation One Dose

INTERVENTIONS:
Drug: Cyclophosphamide — Given by IV
  Arms: Cyclophosphamide
Drug: Mesna — Given by IV
  Arms: Mesna
Drug: Filgrastim — Given by IV
  Arms: Filgrastim
Drug: Melphalan — Given by IV
  Arms: Melphalan
Drug: Fludarabine phosphate — Given by IV
  Arms: Fludarabine phosphate
Drug: Tacrolimus — Given by IV
  Arms: Tacrolimus
Drug: Mycophenolate mofetil — Given by IV
  Arms: Mycophenolate mofetil
Drug: Total Body Irradiation One Dose — Given by IV
  Arms: Total Body Irradiation One Dose

SUMMARY:
The goal of this clinical research study is to learn about the safety and effectiveness of giving KDS-1001 in combination with a standard stem cell transplant to patients with acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), or chronic myeloid leukemia (CML). KDS-1001 is a study product created using certain immune cells called natural killer (NK) cells collected from a third-party donor.

DETAILED DESCRIPTION:
Primary Objective

Assess the safety and effectiveness of "off the shelf" third party NK cells in combination with allogeneic SCT in patients with myeloid malignancies.

Secondary Objectives

To assess NK cell related toxicities To estimate the proportion of patients with engraftment/graft failure. To assess the rate of leukemia relapse, disease-free survival (DFS), overall survival (OS), and GVHD-free, Relapse-free survival (GRFS) after transplantation by one year.

To estimate the non-relapse mortality (NRM) at day 100, day 180 and 1 year post-transplant.

To estimate the cumulative incidence of grade 2-4 and grades 3-4 aGVHD at day 100. To assess the rate of chronic GVHD within the first-year post transplantation. To assess rate of BK, CMV, and Adenovirus infections. To assess MRD. To assess immune reconstitution post-transplant

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 18 to 70 years old at the time of enrollment.
2. Patients weighing at least 42 kg
3. Patient with the hematologic malignancies described below, as well as an HLA matched related donor, HLA matched unrelated donor, a haploidentical related donor, or a one antigen mismatched unrelated donor. HLA matching includes HLA A, B, C, and DR-B1.
4. Patients must have one of the following diseases:

   Acute myeloid leukemia (AML):

   a. With one or more high-risk features defined as: (i) Greater than 1 cycle of induction therapy required to achieve remission; (ii) Preceding myelodysplastic syndrome (MDS);

   Presence of FLT3 mutations or internal tandem duplication or other mutations designated as adverse-risk by the ELN Leukemia Net AML Classification (see Appendix 2):

   Adverse:
   * t(6;9)(p23;q34.1); DEK-NUP214
   * t(v;11q23.3); KMT2A rearranged
   * t(9;22)(q34.1;q11.2); BCR-ABL1
   * inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2); GATA2,MECOM(EVI1)
   * -5 or del(5q); -7; -17/abn(17p)
   * Complex karyotype, monosomal karyotype
   * Wild-type NPM1 and FLT3-ITDhigh
   * Mutated RUNX1
   * Mutated ASXL1
   * Mutated TP53 (iv) FAB M6 or M7 classification; (v) Adverse cytogenetics: -5, del 5q, -7, del7q, abnormalities involving 3q, 9q, 11q, 20q, 21q, 17, +8 or complex karyotype [> 3 abnormalities]; or other mutations designated as adverse-risk by the ELN criteria; (vi) Treatment-related AML (vii) Primary induction failure with partial response to therapy who achieve adequate cytoreduction (viii) Aplastic/hypoplastic marrow with or without detectable persistent disease after induction chemotherapy or after salvage chemotherapy.

   (ix) Have minimal residual disease by flow cytometry, FISH, detection of disease related mutations or cytogenetic abnormality after first course of induction chemotherapy (x) Have relapsed after prior allogeneic hematopoietic transplant

   AND

   b. Patients must be in one of the following (i) CR: complete remission, (ii) CRi: CR with incomplete hematologic recovery, or (iii) MLFS: morphological leukemia-free state with less than 5% bone marrow blasts.

   (iv) If not in either of the above i-iii, then may be in either of the following:
   1. Primary induction failure with partial response to therapy who achieve adequate cytoreduction
   2. Aplastic/hypoplastic marrow with or without detectable persistent disease after induction chemotherapy or after salvage chemotherapy

   Myelodysplastic syndromes (MDS):

   a. De novo MDS with intermediate or high-risk IPSS scores, chronic myelomonocytic leukemia (CMML) or treatment-related MDS. Patients with intermediate-1 features should have failed to respond to hypomethylating agent therapy. .

   Patients must have less than 10% bone marrow blasts

   Chronic myeloid leukemia (CML):
   1. Failed to achieve cytogenetic remission or have cytogenetic relapse after treatment with at least 2 tyrosine kinase inhibitors, or
   2. Accelerated phase or blast phase at any time, or
   3. Intolerant of available TKIs
5. Performance score of at least 70% by Karnofsky or 0 to 1 by ECOG.
6. Adequate major non-hematopoietic organ system function as demonstrated by:

   1. Serum creatinine clearance equal or more than 50 ml/min (calculated with Cockcroft-Gault formula).
   2. Bilirubin equal or less than 1.5 mg/dL except for Gilbert's disease. ALT or AST equal or less than 200 U/L for adults. Conjugated (direct) bilirubin less than 2x upper limit of normal.
   3. Left ventricular ejection fraction equal or greater than 45%.
   4. Diffusing capacity for carbon monoxide (DLCO) equal or greater than 60% predicted corrected for hemoglobin.
7. Ability to understand and willingness to sign the written informed consent document.
8. Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the Investigator while on study.

Exclusion criteria:

1. HIV positive; active hepatitis B or C.
2. Uncontrolled infections; PI is the final arbiter of this criterion.
3. Liver cirrhosis.
4. CNS involvement within 3 months prior to the transplant.
5. Positive pregnancy test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
6. Inability to comply with medical therapy or follow-up.
7. Patient with a known history of allergic reactions to any constituents of the product, including a known history of allergic reactions to cellular products or DMSO.
8. Other malignancy/cancer diagnosis with active disease or in remission and <2 years ago, not including nonmelanoma skin cancer
9. Requiring systemic corticosteroids with prednisone dose >10 mg or equivalent.
10. KDS-1001 Donor specific antibodies (dsa) >3000 MFI units or C1q positive

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Ramdial, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Caner Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered in MD Anderson Cancer Center
Groups:
- NK Cell Infusion in Combination With Fludarabine Melphalan and TBI for Participants Undergoing SCT: D-7 to D-6 Melphalan Administration: Patients < age 60 receive melphalan 140 mg/m2 IV split into two doses (70 mg/m2 IV each day).
  Patients age 60-70 receive melphalan 100 mg/m2 IV (infused per package insert) split into two doses (50 mg/m2 IV each day).
  D-7 to D-4 Fludarabine Administration. Fludarabine will be administered at the dose of 40 mg/m2 IV daily for four doses on days -7 to -4.
  D-3 TBI 200 cGy on D-3. D-2 NK cell (KDS-1001) administration D+3 and D+4 Post Transplant D+5 GvHD prophylaxis with Tacrolimus and Mycophenolate Mofetil
Period: Overall Study
Arm/Group | NK Cell Infusion in Combination With Fludarabine Melphalan and TBI for Participants Undergoing SCT
Started | 24
Completed | 21
Not Completed | 3
Not completed — Due to COVID19 | 1
Not completed — Due to Bacteremia | 1
Not completed — Due to viral infection | 1

BASELINE CHARACTERISTICS:
Arm/Group | NK Cell Infusion in Combination With Fludarabine Melphalan and TBI for Participants Undergoing SCT
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Graft Failure
Description: Primary Graft failure is defined as failure to achieve an ANC > 0.5 x 109/L for 3 consecutive days by day 28 post SC infusion, with no evidence of donor derived cells by bone marrow chimerism studies and no evidence of persistent or relapsing disease.
Time Frame: 28 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | NK Cell Infusion in Combination With Fludarabine Melphalan and TBI for Participants Undergoing SCT
Number analyzed (Participants) | 21
Participants | 0

2. Secondary Outcome: Number of Participants Experienced Non-relapsed Mortality at 100 Day Post Transplant
Description: Number of participants died from any cause other than relapse disease.
Time Frame: 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | NK Cell Infusion in Combination With Fludarabine Melphalan and TBI for Participants Undergoing SCT
Number analyzed (Participants) | 21
Participants | 4

3. Secondary Outcome: Number of Participants in Subsequent Transplant Prior to NK Cell Infusions/Stem Cell Transplant
Description: Number participants had prior allogeneic transplants before study enrollment
Time Frame: On the day of study consent
Measure: Count of Participants; unit: Participants
Arm/Group | NK Cell Infusion in Combination With Fludarabine Melphalan and TBI for Participants Undergoing SCT
Number analyzed (Participants) | 21
Participants | 10

ADVERSE EVENTS:
Time Frame: 100 days
Arm/Group | NK Cell Infusion in Combination With Fludarabine Melphalan and TBI for Participants Undergoing SCT
All-Cause Mortality (participants affected / at risk) | 12/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NK Cell Infusion in Combination With Fludarabine Melphalan and TBI for Participants Undergoing SCT (N=21)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bacterial (Infections and infestations) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fungal (Infections and infestations) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Guillain-Barre Syndrome (Nervous system disorders) | 1 (1)
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 1 (1)
Low granulocyte (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Secondary graft failure (Blood and lymphatic system disorders) | 3 (4)
Viral (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NK Cell Infusion in Combination With Fludarabine Melphalan and TBI for Participants Undergoing SCT (N=21)
(Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
ALT increased (Investigations) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
AST increased (Investigations) | 6 (6)
Bacterial (Infections and infestations) | 14 (25)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Creatinine increased (Investigations) | 10 (10)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 14 (15)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ejection fraction decreased (Cardiac disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9)
Fluid overload (General disorders) | 17 (17)
Fungal (Infections and infestations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hemorrhagic Cystitis (Renal and urinary disorders) | 10 (10)
Hemorrhoids (Gastrointestinal disorders) | 7 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4)
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 9 (9)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 6 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (28)
Ocular GvHD (Eye disorders) | 1 (1)
Oral GvHD (Gastrointestinal disorders) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 9 (9)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 12 (16)
T bilirubin increased (Investigations) | 3 (3)
Tachycardia (Cardiac disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 4 (4)
Tremor (Nervous system disorders) | 3 (3)
Viral (Infections and infestations) | 9 (14)
VOD (Hepatobiliary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT05115630/Prot_SAP_001.pdf